CLINICAL TRIAL: NCT06701123
Title: mHealth to Help Pregnant and Postpartum Women in Recovery for Opioid Use Disorder
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201805132; 5R34DA050453 (NIH)
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Opioid Use Disorders
Keywords: Addiction; mhealth; Women; Substance use disorder; intervention
MeSH Terms: conditions — Opioid-Related Disorders; Behavior, Addictive; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention : Control Group Access to uMAT-R but did not engage (No Intervention): No Intervention : Control Group Access to uMAT-R but did not engage
- Experimental : Experimental Group A- Mobile App with Coaching Feature (Experimental): Access to a coached program on uMAT-R App
  Interventions: Device: uMAT-R mobile app with coaching component

INTERVENTIONS:
Device: uMAT-R mobile app with coaching component — uMAT-R recovery mobile app with coaching component
  Arms: Experimental : Experimental Group A- Mobile App with Coaching Feature

SUMMARY:
The opioid epidemic has resulted in widespread detrimental consequences among vulnerable populations in Missouri, especially among pregnant and postpartum women (PPW) with opioid use disorder (OUD). Perinatal use of medication-assisted treatment (MAT) within a comprehensive treatment plan is the current standard of care, however PPW struggling with OUD may underestimate or misjudge its benefits. At the same time, emerging findings signal that mobile health (mHealth) technologies have the potential to support healthier behaviors among individuals with OUD. In this project, we will test the utility of a theoretically-based digital therapeutics tool (uMAT-R) to encourage MAT adherence and treatment retention while considering the unique needs of PPW. In Aim #1, we will conduct four focus groups with PPW with OUD (target users) on the intervention components of uMAT-R, gathering feedback on theory-driven components that are candidates for inclusion in the tool and eliciting suggestions for additional intervention components. In Aim #2, the tool will be beta-tested for technical/navigational issues among 20 participants. In Aim #3, we will conduct a pilot randomized controlled trial (RCT) among adult PPW with OUD (n=60). This RCT is designed to test the feasibility, acceptability, and preliminary efficacy of uMAT-R (n=40) versus a control group (n=20 who receive treatment-as-usual) regarding participants' treatment adherence, sobriety, and improved MAT attitudes, norms, and perceived control. Recruitment for all Aims will occur at a clinic in St. Louis, Missouri that provides perinatal medication-assisted treatment (MAT) and high-risk maternity care to PPW struggling with OUD. Clinically meaningful effect size and attrition estimates will aid in the planning of a larger RCT in which we will test uMAT-R on a larger scale and expand our recruitment to other clinics across Missouri and other states.

This novel technology could be an invaluable tool to assist physicians in the treatment of OUD among PPW.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant or up to 1 year postpartum
2. Receiving treatment at CARE
3. Adult (≥18 years of age)
4. U.S. resident
5. Currently on MAT
6. Fluent in English
7. women with opioid use disorder (OUD)

   Exclusion Criteria:
8. Currently incarcerated
9. Patients with acute suicidality or psychotic disorders as assessed by CARE providers

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Sobriety | Baseline, 1 month, 2 months, 6 months
  DSM 5 criteria for OUD will be assessed using items from the NSDUH that are based on DSM IV criteria and match all but one of the DSM 5 criteria (craving). Craving will be assessed using the Penn Alcohol Craving Scale (PACS) modified for opioid use.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided